CLINICAL TRIAL: NCT03898661
Title: Local Injection of Collagenase Clostridium Histolyticum (XiapexR) for Refractory Iatrogenic Esophageal Strictures: an Open-label Pilot Study
Brief Title: Collagenase Clostridium Histolyticum for Refractory Iatrogenic Esophageal Strictures
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: unexpected serious adverse event
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGO/2018/004
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Stricture; Esophageal Stricture; Anastomotic; Collagenosis
Keywords: Xiapex; esophageal stricture; stricture; collagenase; refractory; anastomotic
MeSH Terms: conditions — Constriction, Pathologic; Esophageal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- local collagenase (Experimental): Patients receiving local injection of collagenase (0.9 mg XiapexR) into the esophageals stricture
  Interventions: Drug: Collagenase histiolyticum

INTERVENTIONS:
Drug: Collagenase histiolyticum — local injection of collagenase histiolyticum into the esophageal stricture, 1 day before balloon dilation

SUMMARY:
In this open-label pilot study we want to investigate whether intralaesional injection with collagenase clostridium histolyticum (XiapexR) into the esophageal stricture followed by dilation 24 hours later improves the outcome of patients with refractory esophageal anastomotic strictures as compared to dilation alone (standard of care).

DETAILED DESCRIPTION:
Local injection of collagenase clostridium histolyticum (XiapexR) for refractory iatrogenic esophageal strictures: an open-label pilot study.

1. Objective of the study

   To investigate whether intralaesional injection with collagenase clostridium histolyticum (XiapexR) into the esophageal stricture followed by dilation 24 hours later improves the outcome of patients with refractory esophageal anastomotic strictures as compared to dilation alone (standard of care).
2. End point(s) and timepoint(s) of evaluation

Primary outcome measure:

Number of repeat dilations that are required over a timespan of 6 months.

Secondary outcome measures:

1. time to first repeat dilation
2. complication rate.
3. Dysphagia score (0: no dysphagia, able to eat normal diet; 1: moderate passage: able to eat some solid foods; 2: poor passage: able to eat semi-solid foods only; 3: very poor passage: able to swallow liquids only; 4: no passage: unable to swallow anything) 5 General information

3.1 Investigator(s)

Prof Dr. Pieter Hindryckx Department of Gastro-Enterology Ghent University Hospital Pieter.Hindryckx@uzgent.be (+3293320726)

Prof Dr. Danny De Looze Department of Gastro-Enterology Ghent University Hospital Danny.delooze@uzgent.be

Dr. David Tate Department of Gastro-Enterology Ghent University Hospital David.tate@uzgent.be

3.2 Sponsor

Ghent University Hospital, with a grant of the Belgian Society of Gastrointestinal Endoscopy.

3.3 Departments/laboratories involved in the study

Department of Gastro-enterology Ghent University Hospital, Corneel Heymanslaan 10 9000 Ghent

4 Introduction

The main causes of benign esophageal strictures are inflammatory (reflux disease, eosinophilic esophagitis, caustic…) or iatrogenic (post-irradiation, post endoscopic (sub)mucosal resection, post radiofrequency ablation, anastomotic…). Most esophageal strictures respond well to endoscopic balloon dilation. Nonetheless, more than one third of patients develop recurrent symptoms after dilation within the first year (1).

Especially iatrogenic strictures can be difficult to treat and often require multiple dilation sessions to obtain long-term relief of dysphagia (2, 3). According to the Kochman criteria, a refractory stricture is defined as a cicatricial or fibrotic narrowing of the esophageal luminal diameter resulting in clinical symptoms of dysphagia, with an inability to successfully remediate the anatomic problem to a diameter of at least 14 mm over 5 dilation sessions at two-week intervals (4). A recurrent stricture is defined as a cicatricial or fibrotic narrowing with an inability to maintain a satisfactory luminal diameter for four weeks once the target diameter of 14 mm has been achieved (4). Several options (stenting, intralesional injection of corticosteroids, needle knife incision) have been proposed to manage these strictures, with a varying success rate (5). A significant proportion of patients will finally need self-bougienage or surgery (5).

In conclusion, the treatment of esophageal iatrogenic strictures remains a challenge for clinicians and there is an unmet need for novel approaches to manage the patients suffering from this condition in order to avoid repeated dilations and/or invasive surgery.

XiapexR is a locally injectable collagenase approved for the management of Dupuytren's and Peyronie's disease (6, 7). Xiapex is a mixture of two collagenases, enzymes produced by the bacterium Clostridium histolyticum that dismantle collagen. Approximately 24 hours after local injection, the collagen fibres have lost their strength and can be easily broken by manipulation. This therapy has been a breakthrough in the management of Dupuytren's disease, avoiding surgery in the vast majority of patients (6).

After local injection, the collagenases do not reach the bloodstream in significant amounts and are presumed to largely stay at the point of injection until they are broken down by proteases. As a result, side effects are uncommon and are most often injection site reactions including lymphadenopathy (swollen lymph nodes), itching, pain, oedema, and bleeding (for example in the form of bruises or ecchymoses). Allergic reactions are seen in less than 1% of patients (8).

XiapexR has been proposed as a promising treatment for refractory urethral strictures but has never been evaluated in refractory GI strictures (9).

5 The present study

5.1 Study design

Proof of concept open pilot study with a historical control cohort.

5.2 Medication

5.2.1 Composition and dosing

One vial (0.9mg) xiapex in 3ml dissolvent (also provided by the company) will be divided over 4 quadrants within the fibrotic stricture

5.2.2 Producer

Lonza AG Lonzastrasse 3930 Visp Switzerland

5.2.3 Distributor

Swedish Orphan Biovitrum AB SE-112 76 Stockholm Sweden

5.2.4 Packaging

Xiapex powder is supplied in a clear glass vial (3 ml, type I glass) with rubber stopper, aluminium seal and flip-off cap (polypropylene). Solvent: 3 ml solution supplied in a clear glass vial (5 ml, type I glass) with rubber stopper, aluminium seal and flip-off cap (polypropylene).

5.2.5 Administration way

Intralaesional injection.

5.2.6 Labelling

Xiapex is a commercialized product and the commercially available labelling will be used. A study label will be applied to the medication (not obscuring the original label), with following information:

5.2.7 Storage conditions

Store in a refrigerator (2°C - 8°C). Do not freeze.

5.2.8 Known side effects of the medication

After local injection the collagenases do not reach the bloodstream in significant amounts and are presumed to largely stay at the point of injection until they are broken down by proteases. As a result, side effects are uncommon and are most often injection site reactions including lymphadenopathy (swollen lymph nodes), itching, pain, oedema, and bleeding (for example in the form of bruises or ecchymoses). Allergic reactions are seen in less than 1% of patients Drug accountability

5.2.9 Drug accountability

Drug accountability will be documented.

5.3 The subjects

5.3.1 Number of subjects

Active group: 10 patients presenting with iatrogenic esophageal strictures. Control group: A historical cohort that consists of 40 consecutive patients that received an endoscopic balloon dilation 12-15mm for an iatrogenic anastomotic stricture at our centre.

5.3.2 Inclusion criteria

The patient is 18-90 years old The patient suffers from dysphagia caused by an iatrogenic esophageal stricture The stricture is amenable for endoscopic dilation The patient has undergone at least 1 previous endoscopic dilation for the same stricture The patient has signed the ICF

5.3.3 Exclusion criteria The patient is not fluent in Dutch

5.3.4 Replacement of subjects

Patients that are not able to participate to the study will receive the standard of care, consisting of endoscopic dilations alone. Only 1 intralaesional administration of the study drug is given at the start of the experiment. Early drop-out of the study (before 6 months) will therefore not impact further standard care of the patient.

5.3.5 Restrictions and prohibitions for the subjects

* Patient need fasting for at least 8 hours prior to the gastroscopies
* Patients on anticoagulant medication need to interrupt the treatment according to the recommendations of the treating physician (Prof dr. Pieter Hindryckx or prof dr Danny De Looze)

5.3.6 Possible advantages and risks for the subjects

It is possible that participation to the study will result in less need for repeat dilations for the iatrogenic esophageal strictures (unknown).

Every dilation carries the risk of perforation, even in the most experiences hands. No additional dilations are performed in light of the study. It is unknown whether local injection of the study drug augments the risks of perforation.

Every patient is carefully monitored after dilation (standard of care). Upon clinical suspicion of perforation, a CT scan is performed for confirmation. In case of confirmed perforation, endoscopic stenting is immediately performed to bridge the defect, allowing healing of the defect. The stent can most of the time be removed after 6 weeks. Surgical intervention is seldomly needed.

Side effects of the study drug (XiapexR) are expected to be very limited, as the study drug does not enter the bloodstream in significant amounts and is rapidly degraded in the bloodstream by proteases. Local reactions (bleeding, swelling, inflammation) are theoretically possible. Like all foreign substances, Xiapex can induce allergic reactions but these seem to be very rare (only 1 case described in literature).

6 Procedures

6.1 Procedures

After informed consent, patients with an iatrogenic esophageal stricture will receive a first esophagoscopy with local injection of XiapexR injection into the stricture prior to dilatation. One vial (0.9mg) xiapex in 3ml dissolvent (also provided by the company) will be divided over 4 quadrants within the fibrotic stricture. After 24 hours, a second esophagoscopy will be performed to perform balloon dilation of the stricture 12-15mm (standard of care).

The historical cohort will not undergo any procedures, but their patient file will be reviewed to gain outcome data. ICF will be obtained if the patient is still in follow-up at our department.

6.2 Flowchart

* Between day -7 to day -1: Informed consent
* Day 0: Endoscopy, xiapex injection into the strictures (4 quadrants, 0.75ml or 0.25mg per quadrant)
* Day +1: Endoscopy, CRE balloon dilation 12mm to max 15mm
* Day +2 to month 2: clinical evaluation (by phone) every 2 weeks with a window of 3 days (see above for primary and secondary outcome measures)
* Month 2-month 6: Clinical evaluation (by phone) every 4 weeks with a window of 3 days (see above for primary and secondary outcome measures)

The expected total duration of the trial is 18 months.

7 Randomisation / blinding

Not Applicable, as this is an open label trial.

8 Prior and concomitant therapy

Patients on anticoagulant medication need to interrupt the treatment according to the recommendations of the treating physician (Prof dr. Pieter Hindryckx or prof dr Danny De Looze).

All other prior or concomitant medications are allowed

9 Adverse event reporting

List of abbreviations AE Adverse Event CA Competent Authority EC Ethics Committee SAE Serious Adverse Event SSAR Suspected Serious Adverse Reaction SUSAR Suspected Unexpected Serious Adverse Reaction

Adverse events (AE)

The following information will be recorded:

* nature of adverse event
* date and time of occurrence and disappearance
* intensity: mild, moderate or severe
* frequency: once, continuous or intermittent
* decision regarding study: continuation or withdrawal
* relation to the study medication (see below)

AE's will be recorded from the first drug administration until the end of the trial.

Special attention will be given to those subjects who have discontinued the trial for an AE, or who experienced a severe or a serious AE.

Definitions of Adverse Event (AE) Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

Serious Adverse Avent (SAE)

Any untoward medical occurrence that at any dose:

* results in death
* is life-threatening
* requires inpatient hospitalization or prolongation of existing hospitalization,
* results in persistent or significant disability/incapacity, or
* is a congenital anomaly/birth defect.

Note: Medical and scientific judgment should be exercised in deciding whether expedited reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the outcomes listed in the definition above.

Unexpected adverse event An adverse event, the nature or severity of which is not consistent with the applicable product information (e.g., Investigator's Brochure for an unapproved investigational product or package insert/summary of product characteristics for an approved product).

Life-threatening Any event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe.

Associated with the use of the drug An adverse event is considered associated with the use of the drug if the attribution is possible, probable or definitive.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old
* suffers from dysphagia caused by an iatrogenic esophageal stricture
* the stricture is amenable for endoscopic dilation
* the patient has undergone at least 1 previous endoscopic dilation for the same stricture
* signed the ICF

Exclusion Criteria:

* the patient is not fluent in Dutch

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Number of repeat dilations that are required over a timespan of 6 months. | 6 months

SECONDARY OUTCOMES:
time to first repeat dilation | 6 months
complication rate. | 6 months
Dysphagia score | 6 months
  (0: no dysphagia, able to eat normal diet; 1: moderate passage: able to eat some solid foods; 2: poor passage: able to eat semi-solid foods only; 3: very poor passage: able to swallow liquids only; 4: no passage: unable to swallow anything)

CONTACTS AND LOCATIONS:
Locations (1):
- Hindryckx, Zwijnaarde, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/61/NCT03898661/Prot_SAP_000.pdf